CLINICAL TRIAL: NCT07109856
Title: The Peripheral(-Muscle) Oxygenation and Perfusion Score (POPScore) a New Non-invasive Tool to Predict Elevations in C-reactive Protein Levels in Neonates - a Prospective Phase II Observational Study
Brief Title: The Peripheral(-Muscle) Oxygenation and Perfusion Score as a New Non-invasive Tool to Predict Elevations in C-reactive Protein Levels in Neonates
Acronym: POP-Score
Status: Not yet recruiting | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Christina Wolfsberger, MD, Principal Investigator, Medical University of Graz
Other Study IDs: POP-Score; Ethical board number 1010/2025 (Other: Medical University of Graz)
Record Dates: First submitted 2025-07-31; First posted 2025-08-07 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-07

CONDITIONS: Prematurity, Infections; NIRS; Near Infrared Spectroscopy; Preterm Neonates; Term Infant; Infection; Neonatal Sepsis, Early-Onset
Keywords: NIRS; near-infrared spectroscopy; POP-Score; neonates; preterm neonates
MeSH Terms: conditions — Premature Birth; Infections; Neonatal Sepsis | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational cohort: This cohort includes term and moderate-to-late preterm neonates (birth weight ≥ 2000g) with respiratory distress within the first 6 hours after birth, admitted to the neonatal intensive care unit. All enrolled neonates undergo non-invasive monitoring to assess the predictive value of the POP-Score for identifying elevated CRP (≥20 mg/L) within the first 48 hours after birth. The cohort will also be analyzed to evaluate differences in multi-site NIRS measurements (peripheral muscle, cerebral, intestinal, and flank) between those with and without CRP elevation.
  Interventions: Diagnostic Test: POP-Score Assessment; Device: Near-Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Diagnostic Test: POP-Score Assessment — A non-invasive score calculated within the first 6 hours after birth using peripheral muscle oxygenation (pTOI, measured via near-infrared spectroscopy), heart rate, arterial oxygen saturation (SpO2), systolic blood pressure (SABP), and subcutaneous fat layer thickness. The score is evaluated for its ability to predict C-reactive protein (CRP) levels ≥ 20 mg/L within 48 hours.
Device: Near-Infrared Spectroscopy (NIRS) — NIRS measurements are performed within 6 hours after birth using the NIRO 200NX device at four anatomical sites (forearm, forehead, infraumbilical region, and left flank). Measurements assess peripheral muscle, cerebral, intestinal, and flank oxygenation to identify possible differences in tissue perfusion associated with early inflammation or infection.

SUMMARY:
This is a prospective, single-center Phase II observational study investigating the predictive value of the "Peripheral(-muscle) Oxygenation and Perfusion Score" (POP-Score), a novel non-invasive composite index, for early detection of infection/inflammation in neonates. The POP-Score combines peripheral muscle oxygenation measured via near-infrared spectroscopy (NIRS) with routinely monitored clinical parameters (heart rate, oxygen saturation, systolic blood pressure, and subcutaneous fat thickness). The study aims to determine the optimal cut-off value of the POP-Score measured within the first 6 hours after birth to predict elevated C-reactive protein (CRP ≥20 mg/L) within 48 hours. Additionally, multi-site NIRS measurements (cerebral, peripheral muscle, intestinal, and flank) will be evaluated to assess their association with inflammation. The study includes term and moderate-to-late preterm neonates (birth weight ≥2000g) with respiratory distress, admitted to the neonatal intensive care unit at the Medical University of Graz.

DETAILED DESCRIPTION:
Early identification of neonatal infection and inflammation remains a major challenge in neonatal intensive care, particularly in term and moderate-to-late preterm infants with respiratory distress. Current diagnostic approaches rely heavily on clinical symptoms and laboratory markers, which may be subtle or delayed. This study evaluates the diagnostic potential of a novel, non-invasive scoring system-the Peripheral(-muscle) Oxygenation and Perfusion Score (POP-Score)-in predicting elevated C-reactive protein (CRP) levels (≥20 mg/L) within 48 hours after birth.

The POP-Score integrates near-infrared spectroscopy (NIRS)-based peripheral muscle tissue oxygenation measurements (pTOI) with standard clinical monitoring parameters: arterial oxygen saturation (SpO2), heart rate (HR), systolic arterial blood pressure (SABP), and subcutaneous fat layer thickness (measured by ultrasound). A pilot study demonstrated that a POP-Score >1.00 within 6 hours after birth had high sensitivity (100%) and specificity (87%) in predicting elevated CRP values, suggesting potential for early infection screening.

This is a prospective, single-center, observational Phase II study conducted at the Division of Neonatology, Department of Pediatrics and Adolescent Medicine, Medical University of Graz, Austria. Term and moderate-to-late preterm neonates (birth weight ≥2000g) with respiratory distress and risk factors for infection are eligible. Exclusion criteria include severe congenital anomalies, birth weight <2000g, age >6 hours at time of consent, or umbilical artery pH <7.20.

NIRS measurements will be performed within the first 6 hours after birth at four anatomical sites: peripheral muscle (right forearm), cerebral (left forehead), intestinal (infraumbilical), and flank (left posterior flank at T12-L2). Each site will be measured five times using short-duration sensor reapplications to improve data precision. Concurrently, SpO2 and HR (via pulse oximetry), blood pressure, temperature, and subcutaneous fat thickness (via ultrasound) will be recorded. CRP and other laboratory parameters (including leukocyte count, IT-ratio) will be obtained as part of routine care on the first and second day after birth.

The primary aim is to identify the optimal cut-off level of the POP-Score, calculated within the first 6 hours, to predict CRP ≥20 mg/L within 48 hours. Receiver Operating Characteristic (ROC) analysis will be used, with the area under the curve (AUC) estimated and the optimal cut-off determined via the Youden Index.

Secondary aims include evaluating whether multi-site NIRS measurements (cerebral, peripheral muscle, intestinal, and flank) differ significantly between neonates with CRP ≥20 mg/L and those with CRP <20 mg/L, potentially offering additional early indicators of infection or inflammation.

The target sample size is 93 neonates, assuming a 20% incidence of CRP ≥20 mg/L. This allows estimation of the AUC with a 95% confidence interval and acceptable precision. Data will be analyzed using appropriate statistical tests for categorical and continuous variables. Statistical analyses will be conducted in cooperation with the Institute for Medical Informatics, Statistics, and Documentation, Medical University of Graz.

The POP-Score and multi-site NIRS monitoring offer a potentially powerful, non-invasive approach for early identification of at-risk neonates, enabling earlier intervention and improved outcomes. If validated, this tool may support more accurate and timely clinical decision-making in neonatal intensive care settings.

ELIGIBILITY:
Inclusion Criteria:

* birth weight ≥ 2000 grams
* Signs of respiratory distress at time-point of inclusion (tachypnoea >60/min, grunting, intercostal/subcostal/jugular retractions, nasal flaring, supplemental oxygen or respiratory support)
* Decision to conduct full life support
* Written informed consent obtained within the first 6 hours after birth, before inclusion in the study
* Age < 6 hours

Exclusion Criteria:

* No decision to conduct full life support
* No written informed consent
* Birth weight < 2000 grams
* Age > 6 hours
* Severe congenital malformations,
* Umbilical cord artery pH <7.20

Ages: 0 Hours to 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Term and moderate-to-late preterm neonates (birth weight ≥ 2000 grams) with signs of respiratory distress within the first 6 hours after birth, admitted to the neonatal intensive care unit at the Medical University of Graz. All participants must have a gestational age allowing for clinical stability and must meet inclusion criteria including full life support decision and informed consent obtained within 6 hours of birth.
Sampling Method: Non-Probability Sample
Enrollment: 93 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Optimal Cut-Off Value of the POP-Score to Predict Elevated CRP (≥ 20 mg/L) | Within the first 6 hours after birth (parameters of the POP-Score) and CRP within 48 hours
  Determine the optimal cut-off value of the non-invasive POP-Score (unitless score), measured within the first 6 hours after birth, to predict elevated C-reactive protein (CRP) levels (≥ 20 mg/L) within the first 48 hours after birth in neonates with respiratory distress.

SECONDARY OUTCOMES:
Difference in Peripheral Muscle Tissue Oxygenation by NIRS Between Neonates With and Without Elevated CRP | NIRS within 6 hours after birth; CRP within 48 hours
  Evaluate whether there are significant differences in peripheral muscle tissue oxygenation values measured via near-infrared spectroscopy (NIRS) within the first 6 hours after birth between neonates with elevated CRP levels (≥ 20 mg/L) and those with CRP < 20 mg/L.
  Unit of Measure: % tissue oxygen saturation
Difference in Cerebral Tissue Oxygenation by NIRS Between Neonates With and Without Elevated CRP | NIRS within 6 hours after birth; CRP within 48 hours
  Evaluate whether there are significant differences in cerebral tissue oxygenation values measured via near-infrared spectroscopy (NIRS) within the first 6 hours after birth between neonates with elevated CRP levels (≥ 20 mg/L) and those with CRP < 20 mg/L.
  Unit of Measure: % tissue oxygen saturation
Difference in Intestinal Tissue Oxygenation by NIRS Between Neonates With and Without Elevated CRP | NIRS within 6 hours after birth; CRP within 48 hours
  Evaluate whether there are significant differences in intestinal tissue oxygenation values measured via near-infrared spectroscopy (NIRS) within the first 6 hours after birth between neonates with elevated CRP levels (≥ 20 mg/L) and those with CRP < 20 mg/L.
  Unit of Measure: % tissue oxygen saturation
Difference in Flank Tissue Oxygenation by NIRS Between Neonates With and Without Elevated CRP | NIRS within 6 hours after birth; CRP within 48 hours
  Evaluate whether there are significant differences in flank tissue oxygenation values measured via near-infrared spectroscopy (NIRS) within the first 6 hours after birth between neonates with elevated CRP levels (≥ 20 mg/L) and those with CRP < 20 mg/L.
  Unit of Measure: % tissue oxygen saturation

OTHER OUTCOMES:
Difference in Cerebral Fractional Tissue Oxygen Extraction (cFTOE) Between Neonates With and Without Elevated CRP | FTOE within 6 hours after birth; CRP within 48 hours
  Assess whether there are significant differences in cerebral fractional tissue oxygen extraction (cFTOE) values, derived from near-infrared spectroscopy (NIRS), within the first 6 hours after birth between neonates with elevated CRP levels (≥ 20 mg/L) and those with CRP < 20 mg/L.
  Unit of Measure: Unitless ratio
Difference in Peripheral Muscle Fractional Tissue Oxygen Extraction (pFTOE) Between Neonates With and Without Elevated CRP | FTOE within 6 hours after birth; CRP within 48 hours
  Assess whether there are significant differences in peripheral muscle fractional tissue oxygen extraction (pFTOE) values, derived from NIRS, within the first 6 hours after birth between neonates with elevated CRP levels (≥ 20 mg/L) and those with CRP < 20 mg/L.
  Unit of Measure: Unitless ratio
Difference in Intestinal Fractional Tissue Oxygen Extraction (sFTOE) Between Neonates With and Without Elevated CRP | FTOE within 6 hours after birth; CRP within 48 hours
  Assess whether there are significant differences in intestinal fractional tissue oxygen extraction (sFTOE) values, derived from NIRS, within the first 6 hours after birth between neonates with elevated CRP levels (≥ 20 mg/L) and those with CRP < 20 mg/L.
  Unit of Measure: Unitless ratio
Difference in Flank Fractional Tissue Oxygen Extraction (rFTOE) Between Neonates With and Without Elevated CRP | FTOE within 6 hours after birth; CRP within 48 hours
  Assess whether there are significant differences in flank fractional tissue oxygen extraction (rFTOE) values, derived from NIRS, within the first 6 hours after birth between neonates with elevated CRP levels (≥ 20 mg/L) and those with CRP < 20 mg/L.
  Unit of Measure: Unitless ratio

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Division of Neonatology, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pichler G, Pocivalnik M, Riedl R, Pichler-Stachl E, Zotter H, Muller W, Urlesberger B. C reactive protein: impact on peripheral tissue oxygenation and perfusion in neonates. Arch Dis Child Fetal Neonatal Ed. 2012 Nov;97(6):F444-8. doi: 10.1136/archdischild-2011-300578. Epub 2012 Jan 31. PMID 22294473
- [Background] Nanas S, Gerovasili V, Renieris P, Angelopoulos E, Poriazi M, Kritikos K, Siafaka A, Baraboutis I, Zervakis D, Markaki V, Routsi C, Roussos C. Non-invasive assessment of the microcirculation in critically ill patients. Anaesth Intensive Care. 2009 Sep;37(5):733-9. doi: 10.1177/0310057X0903700516. PMID 19775036
- [Background] Chiesa C, Pellegrini G, Panero A, Osborn JF, Signore F, Assumma M, Pacifico L. C-reactive protein, interleukin-6, and procalcitonin in the immediate postnatal period: influence of illness severity, risk status, antenatal and perinatal complications, and infection. Clin Chem. 2003 Jan;49(1):60-8. doi: 10.1373/49.1.60. PMID 12507961
- [Background] Pichler G, Holler N, Baik-Schneditz N, Schwaberger B, Mileder L, Stadler J, Avian A, Pansy J, Urlesberger B. Avoiding Arterial Hypotension in Preterm Neonates (AHIP)-A Single Center Randomised Controlled Study Investigating Simultaneous Near Infrared Spectroscopy Measurements of Cerebral and Peripheral Regional Tissue Oxygenation and Dedicated Interventions. Front Pediatr. 2018 Feb 1;6:15. doi: 10.3389/fped.2018.00015. eCollection 2018. PMID 29450194
- [Background] Grossauer K, Pichler G, Schmolzer G, Zotter H, Mueller W, Urlesberger B. Comparison of peripheral and cerebral tissue oxygenation index in neonates. Arch Dis Child Fetal Neonatal Ed. 2009 Mar;94(2):F156. doi: 10.1136/adc.2008.146654. No abstract available. PMID 19240298
- [Background] Pichler G, Grossauer K, Klaritsch P, Kutschera J, Zotter H, Muller W, Urlesberger B. Peripheral oxygenation in term neonates. Arch Dis Child Fetal Neonatal Ed. 2007 Jan;92(1):F51-2. doi: 10.1136/adc.2005.089037. PMID 17185431
- [Background] Pichler G, Pocivalnik M, Riedl R, Pichler-Stachl E, Morris N, Zotter H, Muller W, Urlesberger B. 'Multi-associations': predisposed to misinterpretation of peripheral tissue oxygenation and circulation in neonates. Physiol Meas. 2011 Aug;32(8):1025-34. doi: 10.1088/0967-3334/32/8/003. Epub 2011 Jun 7. PMID 21654025
- [Background] Pichler G, Wolf M, Roll C, Weindling MA, Greisen G, Wardle SP, Zaramella P, Naulaers G, Pellicer A, Austin T, Bartocci M, Urlesberger B. Recommendations to increase the validity and comparability of peripheral measurements by near infrared spectroscopy in neonates. 'Round table', section of haematology, oxygen transport and microcirculation, 48th annual meeting of ESPR, Prague 2007. Neonatology. 2008;94(4):320-2. doi: 10.1159/000151655. Epub 2008 Sep 11. PMID 18784432
- [Background] Holler N, Urlesberger B, Mileder L, Baik N, Schwaberger B, Pichler G. Peripheral Muscle Near-Infrared Spectroscopy in Neonates: Ready for Clinical Use? A Systematic Qualitative Review of the Literature. Neonatology. 2015;108(4):233-45. doi: 10.1159/000433515. Epub 2015 Aug 25. PMID 26338668
- [Background] Wolfsberger CH, Hoeller N, Baik-Schneditz N, Schwaberger B, Suppan E, Mileder LP, Avian A, Schlatzer C, Urlesberger B, Pichler G. Reference ranges of peripheral-muscle oxygenation in term neonates delivered by Caesarean section during immediate transition after birth. Acta Paediatr. 2024 Dec;113(12):2582-2589. doi: 10.1111/apa.17376. Epub 2024 Aug 8. PMID 39115093
- [Background] Wolfsberger CH, Holler N, Baik-Schneditz N, Schwaberger B, Suppan E, Mileder L, Avian A, Urlesberger B, Pichler G. Peripheral muscle fractional tissue oxygen extraction in stable term and preterm neonates during the first 24 h after birth. Front Pediatr. 2023 Nov 15;11:1276769. doi: 10.3389/fped.2023.1276769. eCollection 2023. PMID 38034828
- [Background] Pichler G, Binder C, Avian A, Beckenbach E, Schmolzer GM, Urlesberger B. Reference ranges for regional cerebral tissue oxygen saturation and fractional oxygen extraction in neonates during immediate transition after birth. J Pediatr. 2013 Dec;163(6):1558-63. doi: 10.1016/j.jpeds.2013.07.007. Epub 2013 Aug 22. PMID 23972642
- [Background] Naulaers G, Morren G, Van Huffel S, Casaer P, Devlieger H. Cerebral tissue oxygenation index in very premature infants. Arch Dis Child Fetal Neonatal Ed. 2002 Nov;87(3):F189-92. doi: 10.1136/fn.87.3.f189. PMID 12390989
- [Background] Bailey SM, Hendricks-Munoz KD, Mally P. Cerebral, renal, and splanchnic tissue oxygen saturation values in healthy term newborns. Am J Perinatol. 2014 Apr;31(4):339-44. doi: 10.1055/s-0033-1349894. Epub 2013 Jul 19. PMID 23873114
- [Background] Alderliesten T, Dix L, Baerts W, Caicedo A, van Huffel S, Naulaers G, Groenendaal F, van Bel F, Lemmers P. Reference values of regional cerebral oxygen saturation during the first 3 days of life in preterm neonates. Pediatr Res. 2016 Jan;79(1-1):55-64. doi: 10.1038/pr.2015.186. Epub 2015 Sep 21. PMID 26389823
- [Background] Wolfsberger C, Baik-Schneditz N, Schwaberger B, Binder-Heschl C, Nina H, Mileder L, Bruckner M, Avian A, Urlesberger B, Pichler G. Changes in peripheral muscle oxygenation measured with near-infrared spectroscopy in preterm neonates within the first 24 h after birth. Physiol Meas. 2020 Aug 11;41(7):075003. doi: 10.1088/1361-6579/ab998b. PMID 32498045
- [Background] Wolfsberger CH, Hoeller N, Suppan E, Schwaberger B, Urlesberger B, Nakstad B, Pichler G. Peripheral fractional oxygen extraction measured with near-infrared spectroscopy in neonates-A systematic qualitative review. Front Pediatr. 2022 Aug 23;10:940915. doi: 10.3389/fped.2022.940915. eCollection 2022. PMID 36081622
- [Background] Jobsis FF. Noninvasive, infrared monitoring of cerebral and myocardial oxygen sufficiency and circulatory parameters. Science. 1977 Dec 23;198(4323):1264-7. doi: 10.1126/science.929199.